CLINICAL TRIAL: NCT07039188
Title: Clinical Evaluation of the Femiset Device for Perineal Descent in Women - Impact on Stool Evacuation
Brief Title: Clinical Evaluation of the Femiset Device for Perineal Descent in Women
Acronym: FEMISET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Sylvie Van den Broeck, Dr., University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 3975
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Perineal Descent; Obstructed Defecation Syndrome (ODS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Femiset (Experimental)
  Interventions: Device: Use device in home environment

INTERVENTIONS:
Device: Use device in home environment — Patients will use the device in their home environment for four weeks.

SUMMARY:
The University of Antwerp developed a device (Femiset) to alleviate defecation difficulties in women suffering from Descending Perineum Syndrome (DPS). The device allows the patient to apply counterpressure to the site of descent (perineal body) during defecation, thereby correcting the excessive descent of the perineum so that the increase in abdominal pressure during the (attempted) defecation results in the evacuation of the stool from the rectum and anus, rather than a further downward pressure on the already descended perineum.

The aim of the clinical study is to validate the efficacy (improvement in defecation) and safety of Femiset as compared to the standard of care of no support to the perineum through a clinical study on 20 patients. The population to be studied consists of adult women suffering from DPS with symptoms of obstructive defecation. Patients will use the device in their home environment for four weeks. The improvement in defecation as perceived by the patient will be assessed with the Patient Global Impression of Change (PGIC) scale. Secondarily, their ODS symptoms will be assessed prior to the test period and at the end of the test period using the Modified Longo Score for ODS. These scores will be compared to determine if there has been an improvement in ODS symptoms. The safety of the device will be validated based on monitoring the incidence of adverse events during the test period. The study will also explore the usability of the device and how it compares to manual perineal support. The results of the study will determine the product's viability.

ELIGIBILITY:
Inclusion Criteria:

* Woman at birth
* Adult (aged 18+)
* ODS complaints
* MRI has been performed within the past three years and a perineal descent of >4cm on MRI (M-Line) is present
* Functional pelvic floor (no dyssynergia)

Exclusion Criteria:

* Scoring less than 7/24 on the modified Longo Score for ODS
* Need for vaginal splinting
* Severe perineal malformations
* Recent perineal surgery (<6 weeks)
* Recent vaginal delivery (<6 weeks)
* Pregnant or actively trying to conceive
* Known allergy to the material of the investigational device
* Inability to follow instructions or handle the device
* Not able to understand the language of the questionnaires (NL/English)
* Incapable of giving informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy - improvement in defecation | 4 weeks
  PGIC Scale
Safety - incidence of adverse events | 4 weeks
  Absence of any adverse events classified with a device-related causality level higher than "not related", as per MDCG 2020-10/1, and assessed by the PI as severe.

SECONDARY OUTCOMES:
Efficacy - improvement in ODS symptoms | 4 weeks
  Modified Longo Score for ODS